CLINICAL TRIAL: NCT05173961
Title: Pilot Study of Mobile Application Designed to Assist Patients Undergoing Radiation Therapy
Brief Title: A Mobile Application, Oncpatient, to Assist Patients Undergoing Radiation Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21564; NCI-2021-13835 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21564 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-12-27; First posted 2021-12-30 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (oncpatient application, survey) (Experimental): Patients use the oncpatient mobile application over the course of radiation therapy. Patients also complete a survey on the final day of radiation treatment.
  Interventions: Other: Internet-Based Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Internet-Based Intervention — Use oncpatient mobile application
Other: Survey Administration — Complete survey

SUMMARY:
This clinical trial determines how well the oncpatient mobile application work in assisting patients undergoing radiation treatment. Radiation therapy can be complex. The technology, daily treatments, and possible side effects can be confusing to prevent and manage. Traditional radiation patient education includes a large amount of information, including details of treatment logistics, side effect prevention, and management. However, this information is not always readily accessible or memorable through the long course of therapy, and critical details can be missed. Oncpatient is a mobile application intended to be a more convenient and accessible form of patient education and guidance that is readily available to help patients and their caretakers navigate through radiation treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of implementing a mobile application designed to be an educational resource designed for patients undergoing radiation treatment.

SECONDARY OBJECTIVES:

I. To assess patient opinions on the usability and helpfulness of the mobile application in helping them through radiation treatments.

II. To assess satisfaction with the mobile application and radiation treatment. III. To assess opinions on existing or new features for the mobile application to be given to future patients.

OUTLINE:

Patients use the oncpatient mobile application over the course of radiation therapy. Patients also complete a survey on the final day of radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older.
* Can read and speak English and provide informed consent.
* Diagnosed with cancer, any stage, any disease site.
* Must be consented to undergo a course of radiotherapy, starting within one month. No limits on duration of radiation apply. Patients must be consented prior to initiating radiotherapy, however.
* Has regular access to a mobile device.

  * Note: This requirement unfortunately leads to the exclusion of underserved patients who cannot afford to have a mobile device. Given that the goal of this study is to establish feasibility of a mobile application, there are no true alternatives, given that these patients would require access to a mobile device if this app were commercially available. However, for impacted patients, the relevant application and resources will be made available on iPads they can access during treatment and a website they can access on any web-enabled device, to ensure they have access as much as reasonably possible. Future iterations of the application will aim to increase access to the resource however possible, but limitations will always apply due to how the core functionality of the app requires a mobile device.

Exclusion Criteria:

* Less than 18 years old.
* Non-English speaking.
* Inability to operate a mobile device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Completion rate | Up to 1 year
  The percent of patients who indicate in the survey that they were able to download the application and use it at least once during radiation will be defined as the completion rate.

SECONDARY OUTCOMES:
Patient opinions on the usability and helpfulness of the mobile application in helping them through radiation treatments | Up to 1 year
  Survey responses and collected demographic data will be evaluated with descriptive statistics where possible. Free-text responses will be recorded and utilized by the application developers to inform future iterations of the application.
Satisfaction with the mobile application and radiation treatment | Up to 1 year
  Survey responses and collected demographic data will be evaluated with descriptive statistics where possible. Free-text responses will be recorded and utilized by the application developers to inform future iterations of the application.
Opinions on existing or new features for the mobile application to be given to future patients | Up to 1 year
  Survey responses and collected demographic data will be evaluated with descriptive statistics where possible. Free-text responses will be recorded and utilized by the application developers to inform future iterations of the application.

CONTACTS AND LOCATIONS:
Overall Officials: Colton Ladbury, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States